CLINICAL TRIAL: NCT02332265
Title: Pathways Linking Poverty, Food Insecurity, and HIV in Rural Malawi
Brief Title: Evaluation of the Effects of a Structural Economic and Food Security Intervention on HIV Vulnerability in Rural Malawi
Acronym: SAGE4Health
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: CARE Malawi (Unknown); University of Pennsylvania (Other); University of Malawi (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lance Weinhardt, Professor, University of Wisconsin, Milwaukee
Other Study IDs: 144-PRJ51ZT; R01HD055868 (NIH)
Record Dates: First submitted 2014-12-21; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: HIV
Keywords: Food Security; Microfinance; Village Savings and Loans; HIV; Quasi-experimental design; Malawi; Structural intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Program Participant Study SAFE area, control area: Participants from two types of areas of rural central Malawi: traditional authorities (TA) selected by CARE to receive the SAFE program (intervention group) and TAs receiving other unrelated CARE programming (controls).
  Intervention TAs: 598 program participants (398 women, 200 men) were interviewed at baseline and 18- and 36-month follow-ups;
  Control TAs: 301 control households were interviewed at baseline and 18- and 36-month follow-ups
  Interventions: Other: Support to Able-Bodied Vulnerable groups to Achieve Food Security (SAFE)
- Community Impact Study, non-SAFE participants: We conducted random surveys (n = 1002)--501 living in the intervention areas but not directly receiving the SAFE intervention and 501 living in the control areas not receiving the SAFE intervention with a 36-month assessment interval, prior to and after implementation of SAFE. Thus, we examined intervention outcomes both in direct SAFE program participants and their larger communities. We used multilevel modeling to examine mediators and moderators of the effects of SAFE on HIV outcomes at the individual and community levels and determine the ways in which changes in HIV outcomes feed back into economic outcomes and food security at later interviews.
- Qualitative SAFE program participant in-depth interview & FGD: We conducted a qualitative end-of-program evaluation consisting of in-depth interviews with 90 SAFE participants.
  Interventions: Other: Support to Able-Bodied Vulnerable groups to Achieve Food Security (SAFE)

INTERVENTIONS:
Other: Support to Able-Bodied Vulnerable groups to Achieve Food Security (SAFE) — The SAFE program was developed & implemented from Jan. 2008-Dec. 2010 by CARE-Malawi, a country office of CARE International, a large NGO. SAFE participants were selected by CARE-Malawi. SAFE was designed to address intertwined structural issues contributing to HIV susceptibility: food insecurity, poverty, gender inequity and ineffective governance. SAFE was implemented in 3 geographic subdivisions (Njombwa, Kaomba, & Mwase) of Kasungu District, located in west-central Malawi. It was funded primarily by the European Commission & partially by the Austrian Development Cooperation. SAFE had 4 main components: 1) improving farming practices & sustainable agriculture through Farmer Field Schools, 2) increasing access to savings and investment through Village Savings & Loans Groups, 3) building capacity of local governance structures & 4) integrating HIV education & gender empowerment into programs through training & education. Details: http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4082534/.
  Groups: Program Participant Study SAFE area, control area; Qualitative SAFE program participant in-depth interview & FGD

SUMMARY:
The purpose of this study is to evaluate a multilevel economic and food security program (Support to Able-Bodied Vulnerable groups to Achieve Food Security; SAFE) in rural central Malawi as implemented and assigned by CARE-Malawi on HIV vulnerability and other health outcomes.

Hypothesis: HIV vulnerability can be reduced through a coordinated set of locally tailored individual and structural interventions that reduces poverty, reduces food insecurity, strengthens community bonds, and addresses gender inequality.

DETAILED DESCRIPTION:
Purpose:

Poverty and lack of a predictable, stable source of food are two fundamental determinants of ill health, including HIV/AIDS. Conversely, episodes of poor health and death from HIV can disrupt the ability to maintain economic stability in affected households, especially those that rely on subsistence farming. However, little empirical research has examined if, and how, improvements in people's economic status and food security translate into changes in HIV vulnerability.

The purpose of the SAGE4Health study is therefore to evaluate a large-scale economic development program implemented by CARE-Malawi to examine mechanisms and magnitude of impact on economic livelihoods, food security, and health. Specifically, the study aims to examine how socioeconomic changes may affect vulnerability to HIV and other risks that can overwhelm rural households in subsistence environments.

To contextualize the study location, it is important to note that HIV/AIDS, poverty and food insecurity contribute substantially to morbidity and mortality in sub-Saharan Africa. The Republic of Malawi, in southeastern Africa, bears one of the heaviest HIV disease burdens globally. Poverty is endemic in Malawi; more than half of its estimated 15 million people live on less than a dollar a day. Food insecurity, defined as having uncertain or limited access to nutritionally adequate food, or being unable to procure food in socially acceptable ways, is an aggravated problem in Malawi.

To better understand the context of HIV in Malawi, and to determine potential responses, it is important to consider HIV within an ecosocial framework. Moving beyond the conventional focus on proximal factors contributing to HIV vulnerability, like individual risk behaviors, it is essential that interventions address poverty and food insecurity as interrelated distal factors in the HIV pandemic, especially in countries like Malawi. Poverty has been consistently recognized as a risk factor for food insecurity and HIV, and food insecurity a risk factor for poor HIV-related outcomes.

Increasing critique has targeted the limitations of proximally focused HIV prevention interventions and emphasizes the need for the development and assessment of complex, multilayered structural interventions that address root causes and causal pathways linking social, economic, political and environmental factors to HIV risk, and vulnerability in specific contexts.There are significant gaps in knowledge, however, about the development, implementation and evaluation of structural interventions. First, while integration of food security interventions into HIV/AIDS prevention programs is essential to curtail the HIV/AIDS pandemic and improve health and quality of life among those infected in resource-poor settings, the literature has offered little guidance to international policy makers, such as the World Food Programme. To our knowledge, there have been no published intervention studies examining the impact of economic status and food security on HIV outcomes in Malawi.

Second, complex multilevel structural interventions are expensive. Typically, non-governmental organizations (NGOs), or government agencies implement them. The cost and complexity of study designs that would adequately evaluate real-world structural interventions do not align well with the typical NIH-funded randomized control trial (RCT) model; this presumably could explain the dearth of research.

Third, major challenges remain in evaluating the impact of structural interventions. Few NGO interventions are evaluated rigorously to rule out alternative explanations for success. Perhaps most importantly, few NGO program evaluations involve a control group. Further, most structural intervention assessments are limited to either structural variables on which they directly intervene (such as social norms that condone intimate-partner violence or microcredit program use rates) or key HIV health outcomes only. These research gaps in the development, implementation and evaluation of structural interventions limit their wider dissemination and scale-up in resource-poor countries, where services are much needed.

The SAGE4Health longitudinal study represents one of the first attempts to understand the mechanisms and processes through which changes in food security and economic outcomes (i.e., income, household assets, livelihood options) can impact HIV vulnerability (i.e., HIV risk behaviors, malnutrition, HIV infections). It also represents one of the first NIH-funded studies based on an academic-economic development NGO partnership. This type of partnership leverages strengths of NGOs (i.e., their ability to respond quickly to crises and their capacity for large-scale, sustainable development work) and the excellence of HIV/AIDS researchers' rigorous study designs and evaluations. In addition to examining pathways linking distal ecosocial factors to HIV vulnerability, this study will provide important information for understanding the impact of multilevel structural interventions on HIV with the potential for sustainable long-term public health benefits. Finally, this collaboration provides a unique opportunity to conduct a detailed study of a multilevel intervention on a scale unlikely to be supported entirely by NIH research funding; in effect, we use the NIH and NGO program funding to enhance both contributions.

Description:

SAGE4Health is a five-year academic-NGO collaboration evaluating the mechanisms and magnitude of the impact of a multilevel economic and food security program (Support to Able-Bodied Vulnerable groups to Achieve Food Security; SAFE), as implemented by CARE-Malawi.

The study is being conducted in the rural areas of the Kasungu District of central Malawi. Among Malawian adults aged 15-49, approximately 11% live with HIV. In Malawi, 74% of people live below the international poverty line of US$1.25 per day. The Malawi economy is dominated by the agriculture sector, which employs 80% of the population, accounts for 42% of national GDP, supplies 81% of foreign exchange earnings and contributes significantly to national and household food security. Aside from agriculture, Malawi's economy is also highly influenced by foreign aid. Based on the World Bank Africa Development Indicators 2011 Report, the foreign aid accounted for 16.3% of Malawi's GDP in 2009. Given that Malawi's economy receives substantial amounts of assistance, there is great interest from both donors and the Malawian government to understand the types of interventions that effectively create sustainable change in both the health and economic sectors.

(see intervention description for full details of SAFE intervention)

SAGE4Health Sample 1: Longitudinal, quasi-experimental, nonequivalent-control group design. Objective: examine impact of SAFE intervention on economic status, food security, HIV/AIDS vulnerability and other health-related outcomes at the SAFE program participants' level. Sample: Participants (n =598) from three Traditional Authorities (TAs) who received SAFE intervention (intervention group) are compared with 301 participants who live in three other matched TAs (control group, matched on demographics and distance from an urban center) not receiving SAFE. Quantitative data was collected in three waves: Baseline (during year 2009), 18-month, and 36-month follow up.

SAGE4Health Sample 2: Random sample community survey with a cohort sequential design. Objective: check the possible threats (i.e., other external factors such as Malawi's national fertilizer and seed programs that were introduced in the same period as the intervention) to the internal validity of the intervention/evaluation by examining whether the intervention effects were the results of something plausible during the study period, in the larger communities where the intervention was delivered. Sample: 500 randomly selected villages in SAFE TAs that were not direct participants in the SAFE program; 500 control TAs, where the SAFE program had not been implemented. Quantitative data was collected in three waves: Baseline (during year 2009), 18-month, and 36-month follow up.

SAGE4Health Sample 3: Series of in-depth qualitative interviews and focus groups conducted 18 months after enrollment near the end of SAFE program implementation. Objective: understand SAFE participants' experiences in the program, their perceptions of its impact and their perspectives on the phenomena. Sample: 90 individuals participating in both focus group discussions and in-depth interviews.

ELIGIBILITY:
Inclusion criteria:

* [Study 1: Prospective participant sample (intervention) and Study 3: End-of-program implementation qualitative sample] (intervention) Participant household in CARE-Malawi SAFE intervention residing in one of three selected study Traditional Authorities
* [Study 1: Prospective control sample] (control) Non-recipients of CARE-Malawi SAFE intervention residing in one of three matched (on demographics and distance from an urban center) Traditional Authorities
* [Study 2: Cross-sectional community sample] (intervention) Non-participant-household in CARE-Malawi SAFE intervention residing in SAFE intervention Traditional Authority
* [Study 2: Cross-sectional community sample] (control) Non-participant-household in CARE-Malawi SAFE intervention not residing in SAFE intervention Traditional Authority

Exclusion criteria:

-[Study 1, 2, and 3] household located in non-study or non-control area Traditional Authority

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: [Study 1] Random selection of households chosen by CARE-Malawi to participate in SAFE intervention residing in Mwase, Kaomba, or Njombwa Traditional Authorities in Malawi. These households are compared to household not receiving the CARE-Malawi SAFE intervention residing in Lukwa, Kawamba, or Chaima.
  [Study 2] Random selection of households in program TAs (Mwase, Kaomba, or Njombwa) including households not receiving intervention. This sample is compared to a random selection of households residing in non-intervention areas TAs (Lukwa, Kawamba, or Chaima).
  [Study 3] Random selection of individuals participating in SAFE intervention within intervention TAs.
Sampling Method: Non-Probability Sample
Enrollment: 1901 (Actual)
Dates: Start 2009-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in economic status | Change in economic status between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention)
  Change in economic status between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention), as measured by a questionnaire containing questions on sources of livelihood (formal employment/wage labor, ganyu/casual labor, crop farming, livestock farming, trading/selling, etc.); exposure and coping methods to economic crises like major illness, environmental disasters, death of household member, etc.; housing quality like roof type (thatched roof, corrugated metal roof, tile, other), floor type (earth/mud, cement, tile, other), wall type (mud, brick, etc.); household assets like ownership of a hoe, axe, sickle, chemical sprayer, treadle pump, plough, etc. and livestock assets such as cattle, dairy cow, sheep, work oxen, etc.
Change in food security | Change in food security between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention)
  Change in food security between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on self-reported number of months in which a household did not have enough food to meet its family's needs; methods for coping with food shortages (such as engaging in ganyu/casual labor, selling firewood/charcoal, sell livestock, borrow cash/food, etc.); as well as quantitative anthropometric measurements of respondents and all household children under five years
Change in HIV vulnerability | Change in HIV vulnerability between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in HIV vulnerability between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention)as measured by as measured by a questionnaire containing questions on self-reported HIV test results, status, and infection risk perceptions and behaviors

SECONDARY OUTCOMES:
Change in dietary diversity | Change in household dietary diversity between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in household dietary diversity between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on self-reported consumption of cereals, legumes, tubers, vitamin A-rich vegetables, vitamin A-rich fruits, meat, milk, fats, tea, etc.
Change in household perceptions of poverty | Change in household perceptions of poverty between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in household perceptions of poverty between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on respondents' self-categorization of their household wealth status; change in livelihood status across the past year; reasons for change in livelihood status
Change in household access to services | Change in household access to services between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in household access to services between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on existing village institutions and receipt of services from different government ministries and NGO programs
Change in sustainable agriculture practices | Change in sustainable agriculture practices between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in sustainable agricultural practices between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on the use of strategies for soil improvement, crop diversification, seed multiplication, drought-tolerant crops, intercropping, etc.
Change in personal health | Change in personal health between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in personal health between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on the respondents' self-reported health status in general, in comparison to others in the village, health status compared to two years ago, physical limitations, frequency of experiencing pain in the past four weeks, etc.
Change in acute and chronic illness | Change in acute and chronic illness between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  6. Change in acute and chronic illness occurrence and healthcare seeking behavior between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on the household's recent need for treatment, where treatment was sought, etc.; and reports of disabled or chronically ill household members
Change in childbirth experiences | Change in childbirth experiences between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in childbirth experiences between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on the location of birth, major problems experienced by women giving birth (i.e. no transport to clinic, high cost, harsh treatment of staff at the health facility, etc.)
Change in family planning | Change in family planning between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in family planning between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on respondents' use (or non-use) and specific methods of family planning
Change in self-reported STD infections | Change in self-reported STD infections between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in self-reported STD infections between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on respondents' experiencing of symptoms potentially indicative of a sexually transmitted infection, type of infection diagnosed, and treatment of such infections
Change in perceived HIV/AIDS stigma | Change in perceived HIV/AIDS stigma between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in perceived HIV/AIDS stigma between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on respondents' likelihood of keeping a family members' status a secret
Change in self-reported male circumcision prevalence and attitudes | Change in self-reported male circumcision prevalence and attitudes between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in self-reported male circumcision prevalence and attitudes between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions on respondents' knowledge of male circumcision and reported circumcision status
Change in gender power attitudes | Change in gender power attitudes between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in gender power attitudes between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions related to male partner treatment of female partners and intimate partner violence (i.e. does the male partner insist on knowing where you are at all times? Does the male partner push or shove you? Does the male partner hit you with his fist or with something else that could hurt you? Etc.)
Change in community cohesion | Change in community cohesion between baseline (early stages of intervention), 18-month follow-up (end of intervention), 36 month follow-up (post-intervention)
  Change in community cohesion between baseline (early stages of intervention), 18-month follow-up (end of intervention), and 36 month follow-up (post-intervention) as measured by a questionnaire containing questions related to scenarios in which the respondent would perceive a neighbor would contribute time or money to a community cause

CONTACTS AND LOCATIONS:
Overall Officials: Lance Weinhardt, PhD, Principal Investigator — University of Wisconsin, Milwaukee, Zilber School of Public Health
Locations (1):
- CARE International-Malawi, Lilongwe, Malawi

REFERENCES:
- [Background] Weiser SD, Tsai AC, Gupta R, Frongillo EA, Kawuma A, Senkungu J, Hunt PW, Emenyonu NI, Mattson JE, Martin JN, Bangsberg DR. Food insecurity is associated with morbidity and patterns of healthcare utilization among HIV-infected individuals in a resource-poor setting. AIDS. 2012 Jan 2;26(1):67-75. doi: 10.1097/QAD.0b013e32834cad37. PMID 21904186
- [Background] Weinhardt LS, Galvao LW, Mwenyekonde T, Grande KM, Stevens P, Yan AF, Mkandawire-Valhmu L, Masanjala W, Kibicho J, Ngui E, Emer L, Watkins SC. Methods and protocol of a mixed method quasi-experiment to evaluate the effects of a structural economic and food security intervention on HIV vulnerability in rural Malawi: The SAGE4Health Study. Springerplus. 2014 Jun 12;3:296. doi: 10.1186/2193-1801-3-296. eCollection 2014. PMID 25019044
- [Background] Bonell CP, Hargreaves J, Cousens S, Ross D, Hayes R, Petticrew M, Kirkwood BR. Alternatives to randomisation in the evaluation of public health interventions: design challenges and solutions. J Epidemiol Community Health. 2011 Jul;65(7):582-7. doi: 10.1136/jech.2008.082602. Epub 2009 Feb 12. PMID 19213758
- [Background] Gupta GR, Parkhurst JO, Ogden JA, Aggleton P, Mahal A. Structural approaches to HIV prevention. Lancet. 2008 Aug 30;372(9640):764-75. doi: 10.1016/S0140-6736(08)60887-9. Epub 2008 Aug 5. PMID 18687460
- [Background] Krieger N. Epidemiology and the web of causation: has anyone seen the spider? Soc Sci Med. 1994 Oct;39(7):887-903. doi: 10.1016/0277-9536(94)90202-x. PMID 7992123
- [Background] Miller CL, Bangsberg DR, Tuller DM, Senkungu J, Kawuma A, Frongillo EA, Weiser SD. Food insecurity and sexual risk in an HIV endemic community in Uganda. AIDS Behav. 2011 Oct;15(7):1512-9. doi: 10.1007/s10461-010-9693-0. PMID 20405316
- [Background] Mkandawire-Valhmu L, Stevens PE. The critical value of focus group discussions in research with women living with HIV in Malawi. Qual Health Res. 2010 May;20(5):684-96. doi: 10.1177/1049732309354283. Epub 2009 Nov 19. PMID 19926798
- [Background] Pronyk PM, Hargreaves JR, Kim JC, Morison LA, Phetla G, Watts C, Busza J, Porter JD. Effect of a structural intervention for the prevention of intimate-partner violence and HIV in rural South Africa: a cluster randomised trial. Lancet. 2006 Dec 2;368(9551):1973-83. doi: 10.1016/S0140-6736(06)69744-4. PMID 17141704
- [Background] Weinhardt LS, Galvao LW, Stevens PE, Masanjala WH, Bryant C, Ng'ombe T. Broadening research on microfinance and related strategies for HIV prevention: commentary on Dworkin and Blankenship (2009). AIDS Behav. 2009 Jun;13(3):470-3. doi: 10.1007/s10461-009-9561-y. Epub 2009 Apr 11. No abstract available. PMID 19363651
- [Background] Victora CG, Habicht JP, Bryce J. Evidence-based public health: moving beyond randomized trials. Am J Public Health. 2004 Mar;94(3):400-5. doi: 10.2105/ajph.94.3.400. PMID 14998803
- [Background] Sumartojo E. Structural factors in HIV prevention: concepts, examples, and implications for research. AIDS. 2000 Jun;14 Suppl 1:S3-10. doi: 10.1097/00002030-200006001-00002. PMID 10981469
- [Background] Sepulveda J. The 'third wave' of HIV prevention: filling gaps in integrated interventions, knowledge, and funding. Health Aff (Millwood). 2012 Jul;31(7):1545-52. doi: 10.1377/hlthaff.2012.0314. PMID 22778344
- [Background] Pronyk PM, Kim JC, Abramsky T, Phetla G, Hargreaves JR, Morison LA, Watts C, Busza J, Porter JD. A combined microfinance and training intervention can reduce HIV risk behaviour in young female participants. AIDS. 2008 Aug 20;22(13):1659-65. doi: 10.1097/QAD.0b013e328307a040. PMID 18670227
- [Background] Laga M, Rugg D, Peersman G, Ainsworth M. Evaluating HIV prevention effectiveness: the perfect as the enemy of the good. AIDS. 2012 Apr 24;26(7):779-83. doi: 10.1097/QAD.0b013e328351e7fb. PMID 22313952
- [Background] Dworkin SL, Blankenship K. Microfinance and HIV/AIDS prevention: assessing its promise and limitations. AIDS Behav. 2009 Jun;13(3):462-9. doi: 10.1007/s10461-009-9532-3. Epub 2009 Mar 18. PMID 19294500
- [Background] Bonell C, Fletcher A, Morton M, Lorenc T, Moore L. Realist randomised controlled trials: a new approach to evaluating complex public health interventions. Soc Sci Med. 2012 Dec;75(12):2299-306. doi: 10.1016/j.socscimed.2012.08.032. Epub 2012 Sep 7. PMID 22989491
- See also: Improved household resilience to economic shocks: findings from SAGE4Health, a mixed-methods, quasi-experimental, non-equivalent control group effectiveness study of a combined structural intervention in rural central Malawi — https://www.youtube.com/watch?v=gpAqoLIzqYY
- See also: International Focus: The Economics of HIV/AIDS in Malawi. Milwaukee Public Television. — https://www.youtube.com/watch?v=s43opna0ho0